CLINICAL TRIAL: NCT04295239
Title: Non-invasive Monitoring of Cerebral Autoregulation in Perioperative Neonatal Cardiac Surgery
Acronym: NEMOCARD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC19_0413
Record Dates: First submitted 2020-02-27; First posted 2020-03-04 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2022-03

CONDITIONS: Congenital Heart Disease in Children; Extracorporeal Circulation; Complications

STUDY DESIGN:
Intervention Model Description: Monocentric, prospective and pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI (Experimental): Pre-operative AND post-operative MRI
  Interventions: Procedure: MRI

INTERVENTIONS:
Procedure: MRI — Pre and Post operative MRI

SUMMARY:
Cardiac surgery under extracorporeal circulation (ECC) in newborns with congenital heart disease causes significant morbidity and mortality. The perioperative period is a period of major vulnerability implicated in the appearance of these sequelae, and it is therefore essential to monitor brain function during ECC. The quality of cerebral oxygenation in the perioperative period is routinely monitored non-invasively by infra-red spectroscopy, which makes it possible to estimate cerebral tissue oximetry from a surface electrode (NIRS). The association between time spent outside the limits of cerebral autoregulation and the occurrence of perioperative encephalopathy is not known. The purpose of this study is to determine whether disturbances in brain autoregulation during the operative period are associated with the occurrence of postoperative encephalopathy in children operated on for congenital heart disease in the neonatal period. The main objective of the research is to determine the association between time spent outside individually determined cerebral autoregulation limits and the appearance of brain lesions suggestive of low brain output. Secondary objectives will investigate the association between time spent outside autoregulatory limits and the occurrence of postoperative encephalopathy defined by clinical and encephalographic criteria and will study factors predictive of the development of postoperative encephalopathy.

ELIGIBILITY:
Inclusion Criteria:

* Any newborn (0-28 days) with congenital heart disease, hospitalized in the preoperative period at the Nantes University Hospital, for whom a decision is made to perform an operation under extracorporeal circulation, suitable to be transported for an MRI without risk, advice taken from the treating team.

Exclusion Criteria:

* emergency cardiac surgery
* Preoperative extracorporeal assistance
* Preoperative intubation
* Preoperative administration of inotropes
* Pre-operative instability contra-indicating pre-operative MRI
* Dependence on a pace maker contra-indicating MRI Imaging.
* Parental consent refusal
* Non-affiliation to a health security insurance

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2022-02-19 (Actual); Study Completion 2022-02-19 (Actual)

PRIMARY OUTCOMES:
determine the association between time spent outside individually determined cerebral autoregulation limits and the development of brain lesions suggestive of low brain output. | 6 weeks after cardiac surgery
  duration of period outside cerebral autoregulation limits, Number, size and extent of new lesions on post-operative MRI.
  Patients will be classified into 2 categories according to whether or not there are new lesions on MRI.
  The lesions retained will be infarcts, white matter lesions and intraparenchymal hemorrhages, classified according to the Magnetic Resonance Imaging Abnormality Scoring System.

SECONDARY OUTCOMES:
describe association between time spent outside autoregulation limits and the occurrence of postoperative encephalopathy defined by clinical and encephalographic criteria. | 6 weeks after cardiac surgery
  duration of period outside cerebral autoregulation limits, Standardized clinical examination according to Amiel Tison at hospital discharge.
describe predictive factors of postoperative encephalopathy | day 1 (cardiac surgery)
  duration of extra-corporal circulation,
describe predictive factors of postoperative encephalopathy | day 1 (cardiac surgery)
  duration of aortic clamp
describe predictive factors of postoperative encephalopathy | day 1 (cardiac surgery)
  duration of selective cerebral perfusion,
describe predictive factors of postoperative encephalopathy | day 1 (cardiac surgery)
  duration of hypothermia deepness
describe predictive factors of postoperative encephalopathy | day 1 (cardiac surgery)
  duration of critical NIRS
describe predictive factors of postoperative encephalopathy | day 1 (cardiac surgery)
  duration of critical median arterial pression (PAM)

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: No